CLINICAL TRIAL: NCT02551367
Title: Letrozole Versus Clomiphene Citrate for Ovulation Induction in Women With Polycystic Ovary Syndrome
Brief Title: Letrozole Versus Clomiphene Citrate for Ovulation Induction in Women With Poly Cystic Ovary Syndrome ( PCOS )
Acronym: LVCCFOROI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: mostafa gomaa hamid halawa (Other)
Collaborators: Ain Shams Maternity Hospital (Other)
Responsible Party: Sponsor-Investigator, mostafa gomaa hamid halawa, Clinical Professor, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8691
Record Dates: First submitted 2015-09-05; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Anovulation; Polycystic Ovary Syndrome
Keywords: letrozole
MeSH Terms: conditions — Anovulation; Polycystic Ovary Syndrome | interventions — Letrozole; Clomiphene; Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- letrozole (Experimental): patients receive letrozole 2.5 mg twice daily from day 2 to day 6 of the cycle , for 3 consecutive cycles, hcg hormone10.000 iu im injection is given when mature follicle diameter reach 18 mm by trans vaginal ultrasound.
  Interventions: Drug: Letrozole; Drug: hcg hormone
- clomiphene citrate (Active Comparator): patients will receive clomiphene citrate 50 mg twice daily from day 2 to day 6 of the cycle for 3 consecutive cycles , hcg 10.000 hormone iu im injection is given when mature follicle diameter reach 18 mm by trans vaginal ultrasound .
  Interventions: Drug: Clomiphene citrate; Drug: hcg hormone

INTERVENTIONS:
Drug: Letrozole — 2.5 mg will taken from day 2 to day 6 of the cycle , for 3 consecutive cycles
  Other Names: femara
  Arms: letrozole
Drug: Clomiphene citrate — 50 mg twice daily orally from day 2 to day 6 , for 3 consecutive cycles
  Other Names: clomid
  Arms: clomiphene citrate
Drug: hcg hormone — 10.000 iu im injection when follicle diameter reach 18 mm by transvaginal ultrasound
  Other Names: pregnyl

SUMMARY:
110 infertile women diagnosed as polycystic ovary syndrome (PCOS) at the age group of 20-35 distributed randomly :

* 55 women will receive letrozole 2.5mg twice daily orally from the 2nd day to the 6thday of the cycle for three successive cycles.
* 55 women will receive clomiphene citrate 50 mg twice daily orally from the 2nd day to the 6thday of the cycle for three successive cycles.

Patients will be subjected to:

Complete history taking:

1. Details about name, age
2. Menstrual history with determination of menarche
3. Amenorrhea or oligomenorrhea , Regularity of the cycle
4. History of endocrine disease.
5. History of previous operations.

   * Physical examination:
   * General examination:

   With special concern to:

   --Acne.

   --Hirsutism .

   --Weight.

   --Height

   --BMI was determined :

   Wt. in kg ـــــــــــــــــــ =

   ) Height in m)2

   - Abdominal examination :
   * for scar of previous pelvic or abdominal operations .

     * Pelvic examination :
   * vaginal examination for enlarged cystic ovaries.

     * ultrasound for diagnosis of pcos.

   PARAMETERS:

(1) rate of ovulation (primary parameter). (2) serum progesterone level on day 21. (3) number of mature follicles produced per cycle. (4) mean endometrial thickness. (6) chemical pregnancy. (7) ongoing pregnancy

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of letrozole on ovulation induction to that of clomiphene citrate in women suffering polycystic ovary syndrome.

Research question:

In women with PCOS , dose letrozole effective in ovulation induction as clomiphene citrate?

Researcher hypothesis:

In women with pcos , letrozole may be as effective as clomiphene citrate in ovulation induction.

Patients and methods Site: this study will be recruited from women attending infertility outpatient clinic at Ain Shams university maternity hospital.

Design: Randomized controlled trial.

Study population: 110 infertile women diagnosed as polycystic ovary syndrome (PCOS) at the age group of 20-35 distributed randomly:

* 55 women will receive letrozole 2.5mg twice daily orally from the 2nd day to the 6thday of the cycle for three successive cycles.
* 55 women will receive clomiphene citrate 50 mg twice daily orally from the 2nd day to the 6thday of the cycle for three successive cycles.

Inclusion criteria:

1. Age between 20-35
2. Primary or secondary infertility
3. Patients diagnosed as PCOS according to Rotterdam criteria :

Menstrual irregularities:

* oligomenorrhea and/or anovulation.
* Oligomenorrhea (menses that occur at intervals greater than 35 days)
* Excess androgen activity. - Clinically: hirsutism .

  * Biochemically: elevated serum androgen. polycystic ovaries (by gynecologic ultrasound)

Exclusion criteria:

Any patients have any causes of infertility other than which mentioned in the inclusion criteria as:

1. Hyperprolactinemia.
2. Male factor of infertility.

   WHO Guidelines 2010 for Normal seminal fluid analysis :

   - Volume> 1.5 ml

   - ph 7.2 to 8.0
   * Liquefaction time 20 to 30 min
   * Sperms concentration >15 million/ml
   * Total motility 40%(Progressive motility + non progressive motility)
   * Progressive motility 32%
   * Morphology > 4% normal forms
3. Thyroid dysfunction.
4. Diabetes Mellitus.
5. Known or suspicious tubal factor infertility ( by hysteroslapingograrhy (HSG) or laparoscope.
6. Endometrioses or pelvic inflammatory diseases .

Patients will be subjected to:

Complete history taking:

1. Details a bout name, age
2. Menstrual history with determination of menarche
3. Amenorrhea or oligomenorrhea , Regularity of the cycle
4. History of endocrine disease.
5. History of previous operations.

   Physical examination:

   General examination:

   With special concern to:

   --Acne.

   --Hirsutism .
   * Weight.
   * Height
   * BMI was determined :

   Wt. in kg ـــــــــــــــــــ =

   ) Height in m)2
   * Abdominal examination:

   for scar of previous pelvic or abdominal operations .
   * Pelvic examination:

   vaginal examination for enlarged cystic ovaries.
   * ultrasound for diagnosis of pcos.
   * The patients will randomly assigned to receive either letrozole (2.5 mg twice daily ) or clomiphene citrate (50 mg twice daily ) from day 2 to day 6 of menstrual cycle .
   * Follicular monitoring will be done by transvaginal ultrasonography (TVS) on alternate days from day 9 of menstrual cycle until a mature follicle detected. Follicle considered mature when it attained 18 mm in size or more by averaging inner two diameters of the follicle.
   * A single injection of 10,000 IU human chorionic gonadotrophin (hCG) will be given, if at least one follicle attained 18 mm. TVS will be done after 48 h of hCG injection to determine follicle rupture. If the follicle found unruptured, TVS repeated after 72 h of the hCG injection to detect whether follicle has ruptured or not. Ovulation ascertained by observing rupture of the follicle by ultrasonogram (USG).
   * Endometrial thickness of 8 mm considered a satisfactory response of the endometrium.
   * on day 21 serum progesterone level will measured. A progesterone level of 10 ng/ml considered as ovulatory.

   PARAMETERS

   Primary outcome measure :

(1) Rate of ovulation assessed by number of mature follicles produced per cycle .

Secondary outcome measures :

(2) Serum progesterone level on day 21 ( assessed up to 24 weeks). (3) Mean endometrial thickness ( assessed up to 24 weeks). (4) Chemical pregnancy ( assessed up to 24 weeks). (5) Ongoing pregnancy ( assessed up to 24 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-35
2. Primary or secondary infertility
3. Patients diagnosed as PCOs according to Rotterdam criteria (Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group.,2003)

Exclusion Criteria:

Any patients have any causes of infertility other than which mentioned in the inclusion criteria as:

1. Hyperprolactinemia.
2. Male factor of infertility.

   WHO Guidelines 2010 for Normal seminal fluid analysis :
   * Volume> 1.5 ml
   * ph 7.2 to 8.0
   * Liquefaction time 20 to 30 min
   * Sperms concentration >15 million/ml
   * Total motility 40%(Progressive motility + non progressive motility)
   * Progressive motility 32%
   * Morphology > 4% normal forms
3. Thyroid dysfunction.
4. Diabetes Mellitus.
5. Known or suspicious tubal factor infertility by HSG or laparoscope.
6. Endometrioses or pelvic inflammatory diseases .

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
ovulation rate | up to 24 weeks.
  Follicular monitoring will be done by transvaginal ultrasonography (TVS) on alternate days from day 9 of menstrual cycle until a mature follicle detected. Follicle considered mature when it attained 18 mm in size or more by averaging inner two diameters of the follicle.
  * A single injection of 10,000 IU hCGwill be given, if at least one follicle attained 18 mm. TVS will be done after 48 h of hCG injection to determine follicle rupture. If the follicle found unruptured, TVS repeated after 72 h of the hCG injection to detect whether follicle has ruptured or not. Ovulation ascertained by observing rupture of the follicle by ultrasonogram (USG).
  * Endometrial thickness of 8 mm considered a satisfactory response of the endometrium.
  * on day 21 serum progesterone level will measured. A progesterone level of 10 ng/ml considered as ovulatory.
  * Ovulation rate is assessed by number of mature follicle (diameter 18-22 mm) per cycle .

SECONDARY OUTCOMES:
day 21 progesterone level | up to 24 weeks
  day 21 serum progesterone level 10 ng/ml is ovulatory
Endomertial thickness | up to 24 weeks
  Endometrial thickness of 8 mm considered a satisfactory response of the endometrium.
On gowing pregnancy | up to 24 weeks
  pregnancy when diagnosed by ultrasound .
Chemical pregnancy | up to 24 weeks
  pregnancy when diagnosed by serum positive hcg test .

CONTACTS AND LOCATIONS:
Overall Officials: mohamed osama, md, Study Director — ain-shams university , cairo